CLINICAL TRIAL: NCT00656396
Title: Does Point of Care Coagulation Testing Reduce the Transfusion of Non-erythrocyte Blood Products in Patients Undergoing Major Surgery? A Randomized-Controlled Trial
Brief Title: Point of Care Coagulation Testing in Patients Undergoing Major Surgery
Acronym: POC-OP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Dr. med. Natalie Urwyler, Departement for Anaesthesiology and Pain Therapy, University Hospital of Bern
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: KEK 232_06; 232_06 (Other: KEK); 3200B0_122461 (Other Grant/Funding Number: SNF); 1295 (Other: Inselspital)
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Blood Loss, Surgical
Keywords: Blood loss; Point of care monitoring; FFP; Major surgery; Prothrombin Time; Blood coagulation tests
MeSH Terms: conditions — Blood Loss, Surgical; Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Standard care
  Interventions: Procedure: Control Intervention
- Intervention (Experimental): Point of care monitoring used
  Interventions: Device: Coagucheck XS Plus (Point of care monitor of coagulation intraoperative)

INTERVENTIONS:
Device: Coagucheck XS Plus (Point of care monitor of coagulation intraoperative) — Coagucheck XS Plus® is used for intraoperative measurement of Prothrombin time
  Other Names: Coagucheck XS Plus® Roche Diagnostics, Basel, Switzerland
  Arms: Intervention
Procedure: Control Intervention — Standard care
  Arms: Control

SUMMARY:
Bleeding is a frequent complication during surgery. The peri-operative administration of blood products, including packed red blood cells, thrombocytes and fresh frozen plasma (FFP), is often deemed necessary. Therefore the transfusion of allogenic blood products mandates strategies to optimize the clinical decision to transfuse. The decision to administer FFP is usually made in the absence of any data. Point of care testing of prothrombin time ensures that a major parameter of coagulation is readily available. The test is fast, easy to perform, inexpensive and may enable physicians to rationally determine the need for FFP. Objective of the study is to determine the effectiveness of point of care coagulation testing of prothrombin time to reduce the administration of FFP.

DETAILED DESCRIPTION:
Background: Bleeding is a frequent complication during surgery. The peri-operative administration of blood products, including packed red blood cells, thrombocytes and fresh frozen plasma (FFP), is often deemed necessary. Beside the expenses of blood products these products carry risks of infection, allergic reaction and immune-modulation. Therefore the transfusion of allogenic blood products mandates strategies to optimize the clinical decision to transfuse. Bleeding during surgery is a dynamic process; it can happen within minutes and result not only in major blood loss, but also in coagulation aberrations. The indication for a transfusion should be based on reliable coagulation studies. Traditional coagulation studies require up to 1 hour. Therefore, the decision to administer FFP is usually made in the absence of any data. Point of care testing of prothrombin time ensures that a major parameter of coagulation is readily available in the operation theatre within 3 minutes. It is fast, easy to perform, inexpensive and may enable physicians to rationally determine the need for FFP. Objective: To determine the effectiveness of point of care coagulation testing of prothrombin time to reduce the administration of FFP. Methods: Patient and assessor blind, single center randomized controlled parallel group trial in 220 patients aged between 18 and 90 years undergoing major surgery (any type, except cardiac surgery and liver transplant) with an estimated blood loss during surgery exceeding 20% of the calculated normal total blood volume or a requirement of FFP according to the judgment of treating surgeons or anesthesiologists. Patients will be randomized to usual care plus point of care coagulation testing or usual care alone without point of care testing. Primary endpoint will be the relative risk to receive any FFP peri-operatively. Significance: Point of care coagulation testing in the operation theatre may reduce the administration of fresh frozen plasma considerably, which in turn may decrease costs and complications usually associated with the administration of allogenic blood products.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 90 years
* Major surgery
* Estimated blood loss during surgery > 20% of individual blood volume of 70ml per kg body weight
* Patients requiring FFP

Exclusion Criteria:

* Known hereditary coagulopathy
* Liver transplant
* Cardiac surgery
* Pregnancy
* Preoperative hemoglobin <100g/l
* Abnormal coagulation studies before surgery
* Active treatment with drugs inhibiting coagulation or platelet function

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2008-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The relative risk to receive any FFP peri-operatively. | at post-operative discharge from hospital, estimated to be about 5 days after randomisation

SECONDARY OUTCOMES:
Number of units of FFP received between randomization and post-operative discharge from hospital | at post-operative discharge from hospital, estimated to be about 5 days after randomisation
The relative risk of major in-hospital bleeding defined as bleeding event requiring an extension of hospitalization, reoperation due to bleeding, bleeding resulting in hemorrhagic shock or death | at post-operative discharge from hospital, estimated to be about 5 days after randomisation
The relative risk of an APTC event (non-fatal myocardial infarction, non-fatal stroke, cardiovascular death, or death of unknown cause) between randomization and post-operative discharge from hospital | at post-operative discharge from hospital, estimated to be about 5 days after randomisation
The relative risk of overall mortality between randomization and post-operative discharge from hospital | at post-operative discharge from hospital, estimated to be about 5 days after randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Robert Greif, MD MME, Study Director — Departement of Anesthesiology and Pain Therapy, Bern University Hospital; Natalie Urwyler, MD, Principal Investigator — Bern University Hospital; Peter Jüni, PD Dr med, Study Chair — CTU Bern, Bern University Hospital, and Institute of Social and Preventive Medicine, University of Bern
Locations (1):
- University Hospital Bern, Bern, Switzerland

REFERENCES:
- [Derived] Urwyler N, Trelle S, Theiler L, Juni P, Staub LP, Luyet C, Alberio L, Stricker K, Greif R. Does point of care prothrombin time measurement reduce the transfusion of fresh frozen plasma in patients undergoing major surgery? The POC-OP randomized-controlled trial. Trials. 2009 Nov 23;10:107. doi: 10.1186/1745-6215-10-107. PMID 19930626